CLINICAL TRIAL: NCT01911247
Title: Preoperative Window Study of Metformin for the Treatment of Endometrial Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1102; 1K23CA143154-01A1 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 850 mg once daily

SUMMARY:
The overall goal of this proposal is to investigate the potential benefit of metformin as a novel therapy for the treatment of endometrial cancer. Investigators will evaluate the effect of short-term metformin treatment on the endometrium of obese women with endometrial cancer by comparing each patient's endometrial biopsy before treatment with metformin to their post-treatment hysterectomy specimen.

Participants: Obese women who are to undergo surgical staging for endometrial cancer will also receive short-term treatment (1-4 weeks) with metformin that will continue until the day prior to surgical staging.

The effect of metformin on proliferation, apoptosis and downstream signaling pathways will be compared between pre-treatment endometrial biopsies and post-treatment hysterectomy specimens. Tissue microarrays will be constructed and immunohistochemstry performed to evaluate proliferation, apoptosis and changes in critical signaling pathways mediated by metformin, and these findings will be correlated with our in vitro preclinical studies. Fresh tissue will also be obtained, and Western immunoblotting will be used to assess expression of the phosphorylated forms of the downstream targets of metformin. The hypothesis is that treatment with metformin will result in a decrease in proliferative markers and an increase in markers of apoptosis in the endometrial cancer tumors. AMPK phosphorylation and inhibition of critical downstream targets of the mTOR pathway will be seen in the post-treatment hysterectomy specimens. Metabolomic profiling will also be performed of tumors and associated biofluids (i.e. serum and urine) before and after treatment with metformin to identify potential biomarkers of response to this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-75 years old
* Have a confirmed diagnosis of type I endometrial cancer (endometrioid) based on pre-operative endometrial biopsy or dilation and curettage (D&C)
* Be obese (BMI greater than or equal to 30) with or without diabetes
* Have no contraindications to short-term metformin therapy
* Have a serum creatinine greater 1.0 mg/dL
* Have normal serum transaminase values (AST and ALT)
* Need to be able to undergo metformin treatment for a minimum of 1 weeks but no more than a maximum of 4 weeks prior to surgical staging

Exclusion Criteria:

* Are currently taking metformin or have taken metformin in the past 6 months or have a history of an allergic reaction or intolerance at any time to metformin
* Have a history of liver or renal dysfunction
* Have a history of alcoholism
* Have a history of vitamin B12 deficiency
* Are pregnant
* Are currently taking insulin
* Are currently taking any hormonal therapy or have been on hormonal therapy in the past 4 weeks
* Are taking a drug that may significantly interact or influence the metabolism of metformin
* In the opinion of the investigator, the patient is felt not to be appropriate for the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in Ki-67 mean levels between pre-metformin treatment endometrial biopsies and post-metformin treatment hysterectomy specimens | 4 weeks
  The primary null hypothesis of interest, that there is no difference between the pre- and post-treatment Ki-67 mean levels will be evaluated using a paired t-test (two-sided, α<0.05 level). Paired t-tests will also be used to compare pre- and post-treatment measures of secondary endpoints. General linear models will be used to explore the relationship between pre-treatment characteristics (e.g., ER, PR, tumor grade) and change in Ki-67, Ki-max and Ki-min.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bae-Jump, M.D. PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Bateman NW, Teng PN, Hope E, Hood BL, Oliver J, Ao W, Zhou M, Wang G, Tommarello D, Wilson K, Litzy T, Conrads KA, Hamilton CA, Darcy KM, Casablanca Y, Maxwell GL, Bae-Jump V, Conrads TP. Jupiter microtubule-associated homolog 1 (JPT1): A predictive and pharmacodynamic biomarker of metformin response in endometrial cancers. Cancer Med. 2020 Feb;9(3):1092-1103. doi: 10.1002/cam4.2729. Epub 2019 Dec 6. PMID 31808620